CLINICAL TRIAL: NCT04529252
Title: Investigating the Genetic and Phenotypic Presentation of Ataxia and Nucleotide Repeat Diseases
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Zbigniew K. Wszolek, Principal Investigator, Mayo Clinic
Other Study IDs: 16-009414
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Spinocerebellar Ataxias; Cerebellar Ataxia; Nucleotide Repeat Disease
MeSH Terms: conditions — Spinocerebellar Ataxias; Cerebellar Ataxia | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Blood draw, we will be collecting up to 100mL (about 7 tablespoons) during the visit.
  * Urine, up to 20 mL of urine will be collected upon proper consent.
  * Stool sample can be collected upon consent.
  * Up to 25 ml (about 5 teaspoons) of CSF will be obtained.
  * Skin biopsy will be obtained using 3 mm skin punch. We will only collect one sample on the patient, but would like to collect an additional skin biopsy on research subjects if the sample is not viable due to technical issues (possible contamination) or because of lack of growth of fibroblasts or there is a need to obtain another sample in the future to assess the progression of the disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Spinocerebellar Ataxia and Other Nucleotide Repeat Diseases: Participants with a clinical diagnosis of spinocerebellar ataxia and other nucleotide repeat diseases (not including Huntington's Disease) with or without a genetic mutation and unaffected family members (grandparents, parents, brothers, sisters, cousins, uncles and aunts) who may or may not carry a genetic mutation for the disease.
  Interventions: Other: Specimen collection
- Control Group: Participants with no known medical or family history of inherited neurodegenerative forms of spinocerebellar ataxia or nucleotide repeat diseases (not including Huntington's Disease) and spouses or caregivers of patients with spinocerebellar ataxia and nucleotide repeat diseases (not including Huntington's Disease) will serve as controls in the study.
  Interventions: Other: Specimen collection

INTERVENTIONS:
Other: Specimen collection — Blood, urine, stool, cerebrospinal fluid, and skin biopsy may be collected

SUMMARY:
The purpose of this study is to create a repository for cerebellar ataxia and nucleotide repeat diseases in order to fully investigate the genetic and phenotypic presentations of both.

DETAILED DESCRIPTION:
The investigators are initiating a new program dedicated to the research and study of neurodegenerative forms of spinocerebellar ataxia as well and other nucleotide repeat diseases with the exclusion of Huntington's Disease. The analysis will be conducted to provide better clinical, genetic, and pathological characterizations of neurodegenerative forms of spinocerebellar ataxia. The investigators would like to create a repository for samples on these cases as well as prospective cases who are seen via clinic, support groups, referrals etc. The investigators will perform clinical evaluations utilizing ataxia pertinent scales. The investigators project to expand the present genealogical bank by collecting more specimens and identify more families in the process. All this will be performed in collaboration with basic scientists in order to conduct proper laboratory investigation that will help arrive at a cure for neurodegenerative forms of spinocerebellar ataxia and nucleotide repeat diseases excluding Huntington's Disease .

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years
* We acknowledge that some participants may be unable to consent due to underlying medical conditions; an eligible proxy may provide the informed consent and provide a signature on the designated line.
* Participants with a clinical diagnosis of spinocerebellar ataxia and other nucleotide repeat diseases (not including Huntington's Disease) with or without a genetic mutation and unaffected family members (grandparents, parents, brothers, sisters, cousins, uncles and aunts) who may or may not carry a genetic mutation for the disease.
* Patients with genetic neurodegenerative form of spinocerebellar ataxia and other nucleotide repeat diseases excluding Huntington's Disease who do not have a known family history of genetic neurodegenerative spinocerebellar ataxia.
* Women of childbearing age will be included as they will not be exposed to any harmful substances nor any forms of treatment while in this study.
* Males and females over 18 years of age with no known medical or family history of inherited neurodegenerative forms of spinocerebellar ataxia or nucleotide repeat diseases (not including Huntington's Disease) will be enrolled as controls.
* Spouses and caregivers of patients with spinocerebellar ataxia and nucleotide repeat diseases (not including Huntington's Disease) may serve as controls in the study.

Controls will also be participants interested in the study after having viewed the advertisement displayed here at Mayo Clinic Florida or heard about the study by word of mouth.

Exclusion Criteria:

* Patients that do not want to participate by either checking no on the contact letter or refusing over the phone. This will be recorded in the Progeny system and patients will not be contacted again.
* Allergy to study-related materials including lidocaine or iodine. We will make all efforts to utilize alternative means when obtaining specimens (i.e. using rubbing alcohol and obtaining blood samples instead of skin biopsies).
* Potential subjects will not be excluded based on being minorities.
* Pregnant subjects will not be included in the study.
* We propose to include 1000 subjects in our repository (500 affected plus unaffected and 500 controls patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified through investigator's clinical practice and their relatives, health fairs, as well as support groups. Controls will be recruited from clinical practice (spouses and caregivers), support groups, and interested volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Development of repository | 10 years
  Specimen sample collection to create a repository for genetic neurodegenerative forms of spinocerebellar ataxia and nucleotide repeat diseases not including Huntington's disease

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew K Wszolek, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials